CLINICAL TRIAL: NCT01439594
Title: Pilot Study to Evaluate Optical Frequency Domain Imaging as a Tool for Assessing the Tissue Response to Radiofrequency Ablation
Brief Title: Optical Frequency Domain Imaging (OFDI) Assessment in Radiofrequency Ablation
Acronym: OFDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2008-P000793
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Esophagus; OCT; Imaging; Radiofrequency Ablation; BARRX
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MGH OFDI Imaging (Experimental): OFDI imaging
  Interventions: Device: MGH OFDI Imaging

INTERVENTIONS:
Device: MGH OFDI Imaging — Imaging of Esophagus with OFDI system

SUMMARY:
The goal of this research is to conduct a pilot clinical study to evaluate the potential use of esophageal Optical Frequency Domain Imaging (OFDI) for assessing the success and degree of injury associated with therapeutic radiofrequency ablation techniques.

DETAILED DESCRIPTION:
This is a single center pilot study conducted in 30 patients scheduled for therapeutic intervention. As the purpose of the study is to assess the response of the esophagus to radio frequency (RF) ablation, and the degree of residual Barrett's Esophagus (BE) remaining following treatment, OFDI imaging of study participants will occur prior to the scheduled BARRX RF treatment, and at the standard 3 and 6 month follow-up visits.

Following initial visual surveillance of the esophagus, the study experimental procedure will begin. Imaging will be performed with the OFDI system in 4 longitudinal (~5cm) volumetric segments that are spaced equally circumferentially along the esophagus in a similar fashion to the standard 4-quadrant biopsy protocol.

Each of the 4 OFDI imaging segments will be acquired in less than 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Barrett's esophagus
* Patients undergoing an Esophagogastroduodenoscopy (EGD)
* Patients scheduled for treatment with RF ablation or patients that have had previous BARRX RF ablation
* Patients must be over the age of 18
* Patient must be able to give informed consent
* Women with child bearing potential must have a negative pregnancy test prior to procedure

Exclusion Criteria:

* Patients on oral anticoagulation medications
* Patients with a history of hemostasis disorders
* Patients that are pregnant
* Patients with esophageal strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachusetts General Hospital; Norman Nishioka, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGH OFDI Imaging
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MGH OFDI Imaging
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of OFDI Imaging as Determined by Number of Successful Imaging Sessions
Description: Images will be taken and compared to standard of care biopsy to assess the success and degree of injury associated with radiofrequency ablation techniques. A successful imaging session is defined as any session where the OFDI device was able to take and produce discernible and clear data that is comparable to corresponding biopsy histopathology. It is considered unsuccessful if we were unable to produce OFDI data and/or attain a corresponding biopsy.
Time Frame: During the OFDI imaging session (about 5 minutes)
Population: A total of 17 Participants took place in this study.
Measure: Number; unit: Imaging sessions
Units Other Than Participants: Completed Imaging sessions
Groups:
- Feasibility: Total number of imaging sessions conducted
Arm/Group | Feasibility
Number analyzed (Participants) | 17
Number analyzed (Completed Imaging sessions) | 64
Imaging sessions
  Imaging sessions with successful OFDI imaging | 64
  Imaging session w/ OFDI & corresponding pathology | 29

ADVERSE EVENTS:
Arm/Group | MGH OFDI Imaging
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No